CLINICAL TRIAL: NCT03345615
Title: Standard Versus Intensive Monitoring After Myocardial Infarction Looking for Atrial Fibrillation
Acronym: SIMPL-AF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Jason Andrade, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: H17-01060
Record Dates: First submitted 2017-11-14; First posted 2017-11-17 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2022-08

CONDITIONS: Atrial Fibrillation New Onset; Myocardial Infarction
Keywords: atrial fibrillation; myocardial infarction; intensive monitoring; oral anticoagulation; hospitalization
MeSH Terms: conditions — Myocardial Infarction; Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: 2:1 enrollment into parallel groups (intensive monitoring vs. standard care).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intensive Monitoring (Experimental): 30-day ambulatory cardiac event monitoir
  Interventions: Diagnostic Test: 30-day ambulatory cardiac event monitor
- Standard Care (No Intervention): Standard Care (no supplemental monitoring)

INTERVENTIONS:
Diagnostic Test: 30-day ambulatory cardiac event monitor — SpiderFlash® 30-day ambulatory cardiac event monitoring will be worn upon discharge.
  Arms: Intensive Monitoring

SUMMARY:
After a myocardial infarction (MI), patients discharged home in sinus rhythm may develop AF that is asymptomatic, undetected, and undertreated. Previous studies (CARISMA and ARREST) have demonstrate high rates of new-onset AF recorded on implantable loop recorder (ILR), although the routine implantation of ILRs post-MI remains costly and invasive. The external loop recorder may effectively identify patients with new-onset AF through a validated diagnostic algorithm and targeted monitoring during a high-risk period (immediately after hospital discharge). We will prospectively randomize patients to receive an external loop recorder or standard care, evaluating rates of new-onset AF developing within 30 days after MI.

DETAILED DESCRIPTION:
The SIMPL-AF trial will evaluate the role of intensive monitoring after myocardial infarction, assessing for new-onset AF after hospital discharge. Patients will be randomized to receive intensive monitoring or standard care in a 2:1 distribution. Patients randomized to intensive monitoring will receive a SpiderFlash® monitor, worn for 30-days after discharge and returned for analysis.

The primary objective of this study is to evaluate at the incidence of new-onset AF at 30-days post-MI using an intensive monitoring strategy, compared to standard of care. Secondary objectives include the impact of intensive monitoring on oral anticoagulation rates at 90-days and 1-year after monitoring, and the risk factors for developing new-onset AF, and the variables associated with initiating or withholding anticoagulation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ST-elevation myocardial infarction (STEMI) or Non-ST-elevation myocardial infarction (NSTEMI; Third Universal Definition of MI) with or without PCI. All patients must have troponin elevation.
* No history of AF during hospitalization, at discharge, or pre-existing AF documented on history (i.e. hospital records, previous hospitalization, ECG records).
* No anticoagulation for AF or other indications (i.e. LV thrombus, heart valves, venous thromboembolism/deep venous thrombosis).
* No concomitant disease expected to reduce expected lifespan to <2 yrs.

Exclusion Criteria:

* Patients receiving CABG surgery during this hospitalization or planned cardiac surgery within the next 3 months.
* Patients with spontaneous coronary artery dissection (SCAD), non-atherosclerotic coronary disease (NACAD), and Takotsubo cardiomyopathy are excluded from this study.
* Patients with contraindications to anticoagulation.
* Patients with a chronic skin disorder on the upper torso, or an allergy to medical tape or glue.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of new-onset AF at 30-days post-MI | 30 days
  New-onset AF detected through intensive monitoring or standard care (routine assessment)

SECONDARY OUTCOMES:
Rate of oral anticoagulation | 90 days and 1-year
  Prescription of anticoagulation after intensive monitoring or standard care
AF-related hospitalization | 90 days and 1-year
  Rates of AF-related hospitalization after intensive monitoring or standard care
Composite cardiovascular and hospitalization events | 90 days and 1-year
  All-cause hospitalization, re-infarction, stroke, and death

CONTACTS AND LOCATIONS:
Overall Officials: Jason G Andrade, MD, Principal Investigator — University of British Columbia
Locations (1):
- Vancouver General Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-09-19): https://cdn.clinicaltrials.gov/large-docs/15/NCT03345615/Prot_SAP_000.pdf
  • Informed Consent Form (2017-11-06): https://cdn.clinicaltrials.gov/large-docs/15/NCT03345615/ICF_001.pdf